CLINICAL TRIAL: NCT00760591
Title: Change of Neutrophil Gelatinase-Associated Lipocalin(NGAL) Following Sodium Phosphate Bowel Preparation(Pilot Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Soon Chun Hyang University (Other)
Responsible Party: Dong Cheol Han MD, Soon Chun Hyang University
Other Study IDs: 2008-41
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: Acute Kidney Failure
Keywords: Acute kidney failure; Colonoscopy; Neutrophil gelatinase-associated lipocalin
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Serum, Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
Oral phosphate purgative is the preferred bowel regimen on the basis of better tolerability, cost effectiveness, and efficacy. There are also numerous reports of patients with even previously normal renal function developing acute and chronic kidney disease after use of oral phosphate purgative. Several uncontrolled case reports and case series suggest a potential link between oral phosphate and acute kidney injury and/or chronic kidney disease1. Its use is contraindicated in patients with preexisting renal disease because of the risk for developing acute renal failure, so called acute phosphate nephropathy, or electrolyte disturbance. Since most of the outpatients who are going to undergo a colonoscopy are exposed to this agent, it is important to detect or prevent vulnerable patients. We would seek a sensitive and rapid diagnosis method of acute kidney injury following sodium phosphate bowel preparation. Within a few hours, NGAL mRNA is highly upregulated after kidney injury, such as renal ischemia-reperfusion and cisplatin nephropathy, NGAL induction precedes the elevation of classical markers for kidney damage such as serum creatinine. The investigators will investigate the change of NGAL following sodium phosphate bowel preparation.

ELIGIBILITY:
Exclusion Criteria:

* Who takes ACE-inhibitor, ARB
* Has a renal or heart disease
* Has a serum electrolyte disturbance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18-65 year old volunteers who want to get colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-09

PRIMARY OUTCOMES:
NGAL | Baseline, colonoscopy day, post 1day, post 2 day

CONTACTS AND LOCATIONS:
Locations (1):
- Soon Chun Hyang University Hospital, Seoul, South Korea